CLINICAL TRIAL: NCT01428479
Title: Phase1 Study of GR121167- A Double Blind, Placebo Controlled, Randomized, Dose Ascending, Single and Multiple Dose Study to Investigate the Safety and Pharmacokinetics Following Intravenous Administration of GR121167 in Healthy Japanese Males-
Brief Title: Phase1 Study of GR121167, Single and Multiple Dose Study in Healthy Japanese Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 115070
Record Dates: First submitted 2011-06-23; First posted 2011-09-05 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Treatment Arm A (Experimental): In Arm A subjects will receive 100 mg of GR121167 in Period 1 and 300 mg of GR121167 in Period 2. In Period 3 subject will receive single doses of placebo on Day 1 and multiple doses of placebo from Day 3 to Day 8
  Interventions: Drug: GR121167 Solution; Drug: Placebo
- Treatment Arm B (Experimental): In Arm B subjects will receive 100 mg of GR121167 in Period 1 and placebo in Period 2. In Period 3 subject will receive 600 mg of GR121167 as single dose on Day 1 and multiple doses of GR121167 from Day 3 to Day8
  Interventions: Drug: GR121167 Solution; Drug: Placebo
- Treatment Arm C (Experimental): In Arm C subjects will receive placebo in Period 1, 300 mg of GR121167 in Period 2. In period 3 subject will receive 600 mg of GR121167 single dose on Day 1 and multiple doses from Day 3 to Day 8
  Interventions: Drug: GR121167 Solution; Drug: Placebo

INTERVENTIONS:
Drug: GR121167 Solution — GR121167 solution will be administered intravenously. For 100 mg subject will receive 10 milliliter (mL) of solution, 30 mL for 300 mg and 60 mL for 600 mg
Drug: Placebo — Placebo solution will be administered intravenously.

SUMMARY:
This study is a randomized, double-blind, ascending dose, placebo-controlled, incomplete crossover, single and multiple dose study in healthy Japanese male subjects to assess the pharmacokinetics and safety/tolerability of single and multiple intravenous administration of GR121167. Serial blood samples and pooled urine samples for the determination of GR121167 concentration will be collected and safety assessments will be performed for each treatment period.

The pharmacokinetics and dose proportionality of GR121167 after single intravenous administration of GR121167 at the dose levels of 100 mg, 300 mg and 600 mg will be assessed. In addition, in the final treatment period (600 mg), twice daily intravenous administrations for 5 days will be also conducted and the pharmacokinetics and accumulation will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as defined as being free from clinically significant illness or disease as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, vital sign, laboratory tests and ECG.
2. Japanese healthy male between 20 and 55 years of age inclusive, at the time of signing the informed consent.
3. Body weight >= 50.0 kg and BMI within the range 18.5<= - <25.0 kg/m2 (inclusive).
4. A creatinine clearance >= 80ml/min as determined by Cockcroft-Gault equation:CLcr (mL/min) = (140 - age) * Wt / (72 * Scr). Where age is in years, weight (wt) is in kg, and serum creatinine (Scr) is in units of mg/dl. [Cockcroft, 1976]
5. Non-smoker or ex-smoker having ceased smoking for at least 6 months.
6. AST, ALT, alkaline phosphatase and total bilirubin =< ULN at screening.
7. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

1. A positive test for syphilis, Hepatitis B surface antigen or positive Hepatitis C antibody, HIV antigen /antibody, HTLV-1 at screening
2. A positive pre-study drug screen at screening.
3. History of regular alcohol consumption exceeding, on average, 14 drinks/week for men (1 drink = 5 ounces (150 mL) of wine or 350 mL of beer or 1.5 ounces (45 mL) of 80 proof distilled spirits) within 6 months of screening.
4. The subject had participated in a clinical study or post-marketing study with an investigational or a non-investigational product during the previous 4 months preceding the first dose of study medication of this study
5. The subject planned to concurrently participate in another clinical study or post-marketing study.
6. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study medication.
7. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy excluding pollen allergy without current symptoms.
8. Where participation in the study would result in donation of blood or blood products in excess of 400 mL within 4 month or 200 mL within 2 months.
9. Unwillingness or inability to follow the procedures outlined in the protocol.
10. Consumption of red wine, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
11. Single QTcB >= 450 msec; at screening
12. Subjects with ECG results considered clinically significant by the investigator.
13. Subjects with a personal history of cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes or additional risk factors for torsades de pointes (e.g., heart failure, hypokalemia).
14. Subjects with a family history of sudden cardiac death.
15. Subjects with a supine systolic blood pressure <90mmHg or >140mmHg and/or a supine diastolic blood pressure <55mmHg or >90mmHg and/or systolic blood pressure drop from supine to standing of >30mmHg.
16. History of renal failure or renal dysfunction

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-01-07 (Actual); Primary Completion 2011-04-04 (Actual); Study Completion 2011-04-04 (Actual)

PRIMARY OUTCOMES:
Profile of pharmacokinetics | Pre, 0.5, 0.75, 1, 1.5, 2, 4, 6 ,8 ,10 ,12 ,24 hrs after single dose and 5 days multiple dose, and at the trough during multiple doses
  Cmax, AUC0-inf, AUC0-last, AUC0-12, C12 (Cτ), accumulation ratios (Ro, Rs)
Safety parameters | upto 24 hrs after dose and 7 days after final dose
  vital signs, ECGs, clinical laboratory tests, and adverse events

SECONDARY OUTCOMES:
Profile of urinary pharmacokinetics | 0-4, 4-8, 8-12, 12-24hrs after single dose
  Ae, fe, CLr
Profile of serum pharmacokinetics | Pre, 0.5, 0.75, 1, 1.5, 2, 4, 6 ,8 ,10 ,12 ,24 hrs after single dose and 5 days multiple dose
  AUC0-24, %AUCex, λz, tmax, t1/2, CL, Vz, Vss

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 115070 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/115070?search=study&search_terms=115070#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 115070 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115070 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115070 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115070 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115070 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115070 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register